CLINICAL TRIAL: NCT03138577
Title: Dose-Response Relationships for Hemidiaphragmatic Paresis Following Ultrasound-Guided Supraclavicular Brachial Plexus Blockade
Brief Title: Dose-Response Relationships for Hemidiaphragmatic Paresis Following Ultrasound-Guided Supraclavicular Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1609017547
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Surgery of Right Upper Extremity
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: A modified "3+3" dose escalation design, modeled after Phase I dose-finding trials, was used to define the dose response curve for local anesthetic volume in the supraclavicular block and resulting hemidiaphragmatic paresis in patients undergoing right upper extremity surgery with supraclavicular block as the primary anesthetic. Possible dosing levels of 5, 10, 15, 20, 25, 30, 35 and 40 mL of local anesthetic were pre-specified with a cohort of three subjects per dose. Diaphragm function was determined by a blinded assessor with M-mode tracings of the right diaphragm before and after supraclavicular block. Secondary objectives included the assessment of respiratory function via negative inspiratory force, oxygen saturation and subjective dyspnea, as well as the extent of sensory and motor blockade.
Who Masked: Outcomes Assessor
Masking Description: The physician reviewing the ultrasound images and determining the presence/absence of diaphragm paralysis is masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Dose Cohort 7 (Other): 5 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine Ultrasound Imaging Bedside Negative Inspiratory Force Meter
  Interventions: Diagnostic Test: Ultrasound Imaging; Drug: Supraclavicular Block; Other: Bedside Negative Inspiratory Force Meter
- Dose Cohort 6 (Other): 10 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine Ultrasound Imaging Bedside Negative Inspiratory Force Meter
  Interventions: Diagnostic Test: Ultrasound Imaging; Drug: Supraclavicular Block; Other: Bedside Negative Inspiratory Force Meter
- Dose Cohort 5 (Other): 15 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine Ultrasound Imaging Bedside Negative Inspiratory Force Meter
  Interventions: Diagnostic Test: Ultrasound Imaging; Drug: Supraclavicular Block; Other: Bedside Negative Inspiratory Force Meter
- Dose Cohort 4 (Other): 20 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine Ultrasound Imaging Bedside Negative Inspiratory Force Meter
  Interventions: Diagnostic Test: Ultrasound Imaging; Drug: Supraclavicular Block; Other: Bedside Negative Inspiratory Force Meter
- Dose Cohort 3 (Other): Supraclavicular Block: 25 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine Ultrasound Imaging Bedside Negative Inspiratory Force Meter
  Interventions: Diagnostic Test: Ultrasound Imaging; Drug: Supraclavicular Block; Other: Bedside Negative Inspiratory Force Meter
- Dose Cohort 2 (Other): 30 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine Ultrasound Imaging Bedside Negative Inspiratory Force Meter
  Interventions: Diagnostic Test: Ultrasound Imaging; Drug: Supraclavicular Block; Other: Bedside Negative Inspiratory Force Meter
- Dose Cohort 1 (Other): 35 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine Ultrasound Imaging Bedside Negative Inspiratory Force Meter
  Interventions: Diagnostic Test: Ultrasound Imaging; Drug: Supraclavicular Block; Other: Bedside Negative Inspiratory Force Meter

INTERVENTIONS:
Diagnostic Test: Ultrasound Imaging — M-mode tracings of right diaphragm motion will be made and recorded by a skilled anesthesiologist. Patients will be examined in the supine position and scanned from a low intercostal or subcostal approach using the liver as an acoustic window. Patients will be asked to perform a "voluntary sniff" (VS) test, for which they will be asked to forcefully inhale through the nose in a sniffing position. The above measurement will be performed immediately preceding the brachial plexus blockade, and then at 15 minute and 30 minutes after block.
Drug: Supraclavicular Block — The patient will be positioned supine with the head turned to the contralateral side. The ultrasound will be placed in the supraclavicular fossa, and the skin and subcutaneous tissues will be infiltrated lateral to the probe with 2% lidocaine. The anesthesiologist can redirect the needle and perform additional injections for complete coverage of the brachial plexus. The local anesthetic will be a 2:1 mix of 1.5% mepivacaine and 0.5% bupivacaine.
Other: Bedside Negative Inspiratory Force Meter — A bedside negative inspiratory force (NIF) meter will be used to measure negative inspiratory force prior to the block and 30 minutes after the block.

SUMMARY:
This clinical trial is for subjects undergoing right upper extremity surgery. The aim of the study is to investigate the dose-response relationship between local anesthetic volume and ipsilateral hemidiaphragmatic paresis (HDP) in patients getting ultrasound-guided supraclavicular brachial plexus blocks in a blinded, prospective trial.

DETAILED DESCRIPTION:
With traditional landmark-based or nerve-stimulator techniques, the incidence of HDP following supraclavicular blocks is approximately 50-67%. Ultrasound-guided techniques are thought to enhance precision while reducing the volume of anesthetic used, but even then HDP incidence is nearly 60%. To date, no trials have studied the dose-response relationship between local anesthetic volume and degree of HDP.

Patient Selection

30 eligible patients undergoing right upper extremity surgery and eligible for supraclavicular blocks will be recruited at NewYork-Presbyterian/Weill Cornell Medical Center.

Evaluation of HDP

Baseline M-mode recordings of diaphragm function will be made by an anesthesiologist. Patients will perform "voluntary sniff" (VS) tests, or forceful nasal inhales, immediately preceding the brachial plexus blockade, and again at 15 minutes and 30 minutes after the block.

Diaphragmatic excursion from baseline will be measured in centimeters; three measurements will be made and averaged. Hemidiaphragmatic paresis will be defined as greater than or equal to 60% reduction in diaphragmatic excursion, no movement, or paradoxical movement in the VS test.

Evaluation of Pulmonary Function

A bedside negative inspiratory force (NIF) meter will be used to measure negative inspiratory force prior to the block and 30 minutes after the block.

Evaluation of Supraclavicular Block

At the 15- and 30-minute marks, the investigators will assess sensory blockade and motor block in the axial, musculocutaneous, radial, median, and ulnar distributions. Both will be judged on 3-point scales. The investigators will also apply a 0-10 point verbal rating scale to assess dyspnea at 30 minutes. Oxygen saturation will be measured off of supplemental oxygen before the block and 30 minutes after the block.

Following the assessments, patients will have surgery using brachial plexus blockade as the primary anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing right upper extremity surgery with supraclavicular block as the primary anesthetic
* Age greater than or equal to 18 years of age
* American Society of Anesthesiologists (ASA) physical status 1 to 3
* Able to give informed consent

Exclusion Criteria:

* Patient refusal for supraclavicular block
* Inability to give informed consent
* Allergy to local anesthetics
* Hemidiaphragmatic dysfunction, suspected or known pulmonary disease
* Neuromuscular disease
* Obstructive or restrictive pulmonary disease
* Medical or anatomic contraindication to supraclavicular blockade as judged by clinician
* Pregnancy

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Tedore, MD, Principal Investigator — WCMC, NYP
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renes SH, Spoormans HH, Gielen MJ, Rettig HC, van Geffen GJ. Hemidiaphragmatic paresis can be avoided in ultrasound-guided supraclavicular brachial plexus block. Reg Anesth Pain Med. 2009 Nov-Dec;34(6):595-9. doi: 10.1097/aap.0b013e3181bfbd83. PMID 19916254
- [Background] Petrar SD, Seltenrich ME, Head SJ, Schwarz SK. Hemidiaphragmatic paralysis following ultrasound-guided supraclavicular versus infraclavicular brachial plexus blockade: a randomized clinical trial. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):133-8. doi: 10.1097/AAP.0000000000000215. PMID 25650633
- [Background] Kant A, Gupta PK, Zohar S, Chevret S, Hopkins PM. Application of the continual reassessment method to dose-finding studies in regional anesthesia: an estimate of the ED95 dose for 0.5% bupivacaine for ultrasound-guided supraclavicular block. Anesthesiology. 2013 Jul;119(1):29-35. doi: 10.1097/ALN.0b013e31829764cf. PMID 23648519
- [Background] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Background] Mier-Jedrzejowicz A, Brophy C, Moxham J, Green M. Assessment of diaphragm weakness. Am Rev Respir Dis. 1988 Apr;137(4):877-83. doi: 10.1164/ajrccm/137.4.877. PMID 3354995
- [Background] Soares LG, Brull R, Lai J, Chan VW. Eight ball, corner pocket: the optimal needle position for ultrasound-guided supraclavicular block. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):94-5. doi: 10.1016/j.rapm.2006.10.007. No abstract available. PMID 17196502
- [Background] Tedore TR, YaDeau JT, Maalouf DB, Weiland AJ, Tong-Ngork S, Wukovits B, Paroli L, Urban MK, Zayas VM, Wu A, Gordon MA. Comparison of the transarterial axillary block and the ultrasound-guided infraclavicular block for upper extremity surgery: a prospective randomized trial. Reg Anesth Pain Med. 2009 Jul-Aug;34(4):361-5. doi: 10.1097/AAP.0b013e3181ac9e2d. PMID 19574870
- [Background] O'Quigley J, Pepe M, Fisher L. Continual reassessment method: a practical design for phase 1 clinical trials in cancer. Biometrics. 1990 Mar;46(1):33-48. PMID 2350571
- [Background] Garrett-Mayer E. The continual reassessment method for dose-finding studies: a tutorial. Clin Trials. 2006;3(1):57-71. doi: 10.1191/1740774506cn134oa. PMID 16539090
- [Background] Neal JM. Ultrasound-Guided Regional Anesthesia and Patient Safety: Update of an Evidence-Based Analysis. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):195-204. doi: 10.1097/AAP.0000000000000295. PMID 26695877
- [Derived] Tedore TR, Lin HX, Pryor KO, Tangel VE, Pak DJ, Akerman M, Wellman DS, Oden-Brunson H. Dose-response relationship between local anesthetic volume and hemidiaphragmatic paresis following ultrasound-guided supraclavicular brachial plexus blockade. Reg Anesth Pain Med. 2020 Dec;45(12):979-984. doi: 10.1136/rapm-2020-101728. Epub 2020 Oct 1. PMID 33004656

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited from August 2018 to July 2019. Fifty-nine subjects were assessed for eligibility. Fourteen subjects were excluded or refused to participate, and 21 were eligible but not approached due to the anticipation of insufficient time to complete assessments. Twenty-four patients consented to enrollment.
Pre-assignment Details: 3 of the 24 enrolled patients were excluded due to baseline abnormal diaphragm motion or inability to visualize the diaphragm on baseline ultrasound scan.
Groups:
- Dose Cohort 7: Supraclavicular block performed with 5 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 6: Supraclavicular block performed with 10 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 5: Supraclavicular block performed with 15 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 4: Supraclavicular block performed with 20 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 3: Supraclavicular block performed with 25 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 2: Supraclavicular block performed with 30 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 1: Supraclavicular block performed with 35 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
Period: Overall Study
Arm/Group | Dose Cohort 7 | Dose Cohort 6 | Dose Cohort 5 | Dose Cohort 4 | Dose Cohort 3 | Dose Cohort 2 | Dose Cohort 1
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 5 mL: 5 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- 10 mL: 10 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- 15 mL: 15 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- 20 mL: 20 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- 25 mL: 25 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- 30 mL: 30 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- 35 mL: 35 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Total: Total of all reporting groups
Arm/Group | 5 mL | 10 mL | 15 mL | 20 mL | 25 mL | 30 mL | 35 mL | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 3 | 1 | 2 | 3 | 13
  >=65 years | 2 | 2 | 1 | 0 | 2 | 1 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 20
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
ASA Classification [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) Classification:
  I: Normal, healthy patient II: Patient with mild systemic disease III: Patient with severe systemic disease
  Participants
    ASA Class I | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 5
    ASA Class II | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 15
    ASA Class III | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper Extremity Surgery Location [Count of Participants; unit: Participants]
  Proximal to elbow | 1 | 1 | 2 | 2 | 0 | 1 | 2 | 9
  Mid arm (at elbow) | 2 | 2 | 1 | 1 | 2 | 1 | 0 | 9
  Distal to elbow | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Hemidiaphragmatic Paresis at Various Volumes of Local Anesthetic 15 Minutes After Supraclavicular Block
Description: Diaphragm motion was recorded during voluntary sniffing fifteen minutes after supraclavicular block with the specified volume of local anesthetic. Blinded investigators reviewed the scans and determined whether the scans were indicative of hemidiaphragmatic paresis (HDP) or not (No HDP). This data was fit to a dose response curve.
Time Frame: 15 minutes
Measure: Count of Participants; unit: Participants
Groups:
- Dose Cohort 7 (5 mL): Supraclavicular block performed with 5 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 6 (10 mL): Supraclavicular block performed with 10 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 5 (15 mL): Supraclavicular block performed with 15 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 4 (20 mL): Supraclavicular block performed with 20 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 3 (25 mL): Supraclavicular block performed with 25 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 2 (30 mL): Supraclavicular block performed with 30 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
- Dose Cohort 1 (35 mL): Supraclavicular block performed with 35 mL of 2:1 mixture of 1.5% mepivacaine and 0.5% bupivacaine
Arm/Group | Dose Cohort 7 (5 mL) | Dose Cohort 6 (10 mL) | Dose Cohort 5 (15 mL) | Dose Cohort 4 (20 mL) | Dose Cohort 3 (25 mL) | Dose Cohort 2 (30 mL) | Dose Cohort 1 (35 mL)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3
Participants
  HDP | 1 | 1 | 1 | 2 | 2 | 3 | 3
  No HDP | 2 | 2 | 2 | 1 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Dose Cohort 7 (5 mL) vs Dose Cohort 6 (10 mL) vs Dose Cohort 5 (15 mL) vs Dose Cohort 4 (20 mL) vs Dose Cohort 3 (25 mL) vs Dose Cohort 2 (30 mL) vs Dose Cohort 1 (35 mL); Test type: Other; Counts and percentages of cases with paralysis were calculated separately for each volume of local anesthetic

2. Primary Outcome: Number of Subjects With Hemidiaphragmatic Paresis at Various Volumes of Local Anesthetic 30 Minutes After Supraclavicular Block
Description: Diaphragm motion was recorded during voluntary sniffing 30 minutes after supraclavicular block with the specified volume of local anesthetic. Blinded investigators reviewed the scans and determined whether the scans were indicative of hemidiaphragmatic paresis (HDP) or not (No HDP). This data was fit to a dose response curve.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Cohort 7 (5 mL) | Dose Cohort 6 (10 mL) | Dose Cohort 5 (15 mL) | Dose Cohort 4 (20 mL) | Dose Cohort 3 (25 mL) | Dose Cohort 2 (30 mL) | Dose Cohort 1 (35 mL)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3
Participants
  HDP | 1 | 1 | 1 | 2 | 3 | 3 | 3
  No HDP | 2 | 2 | 2 | 1 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Dose Cohort 7 (5 mL) vs Dose Cohort 6 (10 mL) vs Dose Cohort 5 (15 mL) vs Dose Cohort 4 (20 mL) vs Dose Cohort 3 (25 mL) vs Dose Cohort 2 (30 mL) vs Dose Cohort 1 (35 mL); Test type: Other; Counts and percentages of cases with paralysis were calculated separately for each volume of local anesthetic; Counts and percentages of cases with paralysis were calculated separately for each volume of local anesthetic

3. Secondary Outcome: Change in Negative Inspiratory Force (NIF) at 30 Minutes
Description: The change of the absolute value of NIF from the baseline measurement to that at 30 minutes after the block
Time Frame: 30 minutes
Measure: Median (Inter-Quartile Range); unit: cm H2O
Groups:
- Subjects With HDP: All subjects, regardless of local anesthetic dose, that demonstrated HDP 30 minutes after block placement.
- Subjects Without HDP: All subjects, regardless of local anesthetic dose, that did not demonstrate HDP 30 minutes after block placement.
Arm/Group | Subjects With HDP | Subjects Without HDP
Number analyzed (Participants) | 14 | 7
cm H2O | -7.5 [-22.0 to 0] | 0 [-10 to 0]
Statistical Analysis 1: Comparison: Subjects With HDP; Test type: Other; p = 0.01, Sign test; Median Difference (Final Values) = 7.5
Statistical Analysis 2: Comparison: Subjects Without HDP; Test type: Other; p = 1.00, Sign test; Median Difference (Final Values) = 0

4. Secondary Outcome: Dose Response Curve for Motor and Sensory Block 15 Minutes After Block
Description: As described in the protocol, each subject's block was assessed via motor and sensory exam at 15 minutes and given a score (0-20), with 20 being a perfect block and any score less than 10 indicating an ineffective block. A dose response curve was generated for block score with different volumes of local anesthetic administered.
Time Frame: 15 minutes
Measure: Number; unit: score on a scale
Arm/Group | Dose Cohort 7 (5 mL) | Dose Cohort 6 (10 mL) | Dose Cohort 5 (15 mL) | Dose Cohort 4 (20 mL) | Dose Cohort 3 (25 mL) | Dose Cohort 2 (30 mL) | Dose Cohort 1 (35 mL)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3
score on a scale
  Subject 1/3 | 1 | 11 | 7 | 2 | 20 | 15 | 11
  Subject 2/3 | 12 | 12 | 0 | 1 | 19 | 15 | 15
  Subject 3/3 | 10 | 0 | 18 | 0 | 5 | 16 | 19
Statistical Analysis 1: Comparison: Dose Cohort 7 (5 mL) vs Dose Cohort 6 (10 mL) vs Dose Cohort 5 (15 mL) vs Dose Cohort 4 (20 mL) vs Dose Cohort 3 (25 mL) vs Dose Cohort 2 (30 mL) vs Dose Cohort 1 (35 mL); Test type: Other; Dose response data was fit with a non-parametric smoothing technique for locally weighted regression (lowess) to produce a dose response curve

5. Secondary Outcome: Dose Response Curve for Motor and Sensory Block Score 30 Minutes After Block
Description: As described in the protocol, each subject's block was assessed via motor and sensory exam at 30 minutes and given a score (0-20), with 20 being a perfect block and any score less than 10 indicating an ineffective block. A dose response curve was generated for block score with different volumes of local anesthetic administered.
Time Frame: 30 minutes
Measure: Number; unit: score on a scale
Arm/Group | Dose Cohort 7 (5 mL) | Dose Cohort 6 (10 mL) | Dose Cohort 5 (15 mL) | Dose Cohort 4 (20 mL) | Dose Cohort 3 (25 mL) | Dose Cohort 2 (30 mL) | Dose Cohort 1 (35 mL)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3
score on a scale
  Subject 1 of 3 | 2 | 14 | 8 | 20 | 20 | 14 | 15
  Subject 2 of 3 | 18 | 14 | 2 | 10 | 20 | 16 | 18
  Subject 3 of 3 | 10 | 12 | 18 | 16 | 16 | 16 | 19
Statistical Analysis 1: Comparison: Dose Cohort 7 (5 mL) vs Dose Cohort 6 (10 mL) vs Dose Cohort 5 (15 mL) vs Dose Cohort 4 (20 mL) vs Dose Cohort 3 (25 mL) vs Dose Cohort 2 (30 mL) vs Dose Cohort 1 (35 mL); Test type: Other; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: Change in Room Air Oxygen Saturation at 30 Minutes.
Description: The change in room air oxygen saturation from baseline to 30 minutes after the block was calculated.
Time Frame: 30 minutes
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Subjects With HDP | Subjects Without HDP
Number analyzed (Participants) | 14 | 7
percent | -1 [-2 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Subjects With HDP; Test type: Other; p = 0.01, Sign test; Median Difference (Final Values) = -1
Statistical Analysis 2: Comparison: Subjects Without HDP; Test type: Other; p = 1.00, Sign test; Median Difference (Final Values) = 0

7. Secondary Outcome: Subjective Dyspnea 30 Minutes After Block
Description: 30 minutes after the block, patients were asked to rate any symptoms of dyspnea on a scale of 0 (no trouble breathing) to 10 (extreme trouble breathing).
Time Frame: 30 minutes
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Subjects With HDP | Subjects Without HDP
Number analyzed (Participants) | 14 | 7
score on a scale | 0 [0 to 2] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Subjects With HDP vs Subjects Without HDP; Test type: Other; p = 0.08, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Dose Cohort 7 (5 mL) | Dose Cohort 6 (10 mL) | Dose Cohort 5 (15 mL) | Dose Cohort 4 (20 mL) | Dose Cohort 3 (25 mL) | Dose Cohort 2 (30 mL) | Dose Cohort 1 (35 mL)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
1. The subjects enrolled in this trial were predominantly female.
2. The subject population studied was free from baseline respiratory disease.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT03138577/Prot_SAP_000.pdf